CLINICAL TRIAL: NCT05357352
Title: Effect of Patient Demographics, Comorbidities, and Medications on Severity of NASH Fibrosis
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 002.HEP.2019.D
Record Dates: First submitted 2021-11-09; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis
Keywords: NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NAFLD/NASH — the characteristics of patients with advanced fibrosis in a community-based referral center.
  Other Names: characteristics of patients

SUMMARY:
Few studies have evaluated an extensive list of possible risk factors for NAFLD for their association with presence and severity of histologic features. We wish to conduct a retrospective study on these possible factors (including demographics, comorbid diseases, and medications) for their association, if any, with severity of histopathologic findings. This study hypothesize that certain risk factors, specifically those contributing to or consisting of metabolic syndrome, will have higher NASH Fibrosis stages.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in Western countries, and is projected to become one of the foremost indications for liver transplantation (2). Both NAFLD and its most severe histopathologic subtype, non-alcoholic steatohepatitis (NASH) can progress to cirrhosis and its complications including hepatic malignancy, and are thus an important target for study. It is well-known that several risk factors are associated with the development of NAFLD, including obesity, type 2 diabetes mellitus, and metabolic syndrome (1), however their association with the presence and severity of histologic features of NAFLD/NASH has not been extensively examined. This study can help determine prognostic indicators for NALFD/NASH which can be useful in its prevention and treatment.

This is a retrospective chart review and de-identified data analysis. Data will be extracted from the patient database from the Methodist Liver Institute from April 2013 - June 2020. Patients with confirmed NAFLD/NASH via liver biopsy will be selected and NAFLD Activity Score and Fibrosis stage will be assessed. Data will then be collected on demographics, comorbid diseases, and medications from EPIC EMR system used by Methodist Health System.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified to have biopsy-proven NASH within April 2013 - June 2020
* Minimum age 18, no upper limit of age
* Patients with complete records

Exclusion Criteria:

* Age <18 years
* Incomplete records
* Diseases other than NASH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed NAFLD/NASH via liver biopsy from the patient database from the Methodist Liver Institute from April 2013 - June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
NAS score lover | April 2013 - June 2020
  Severity of Nonalcoholic fatty liver disease and fibrosis staging. The NAS is a measure of grade and is the sum of numerical scores applied to steatosis (0-3), hepatocellular ballooning (0-2), and lobular inflammation (0-3). Accordingly, the NAS ranges from 0 to 8 (see Table 12.3). The NAS is one of the few grading systems for NAFLD that has been externally validated.

CONTACTS AND LOCATIONS:
Overall Officials: Mantry Parvez, MD, Principal Investigator — The Liver Institute at Methodist Dallas Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No